CLINICAL TRIAL: NCT02878083
Title: Development of a Biomarker of Efficacy of Vedolizumab (EnTyvio®) in Patients With ulcErative ColiTis (DETECT)
Acronym: DETECT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the CELLVIZIO device required to analyse biopsy is available until september 2020
Sponsor: Nantes University Hospital (Other)
Collaborators: Takeda (Industry); Mauna Kea Technologies (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC15_0457
Record Dates: First submitted 2016-08-16; First posted 2016-08-25 (Estimated); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: ULCERATIVE COLITIS
Keywords: vedolizumab,; confocal endomicroscopy; biomarker; ULCERATIVE COLITIS
MeSH Terms: conditions — Colitis, Ulcerative | interventions — vedolizumab; Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VEDOLIZUMAB (Experimental): 300 mg IV
  Interventions: Drug: VEDOLIZUMAB; Drug: ADALIMUMAB

INTERVENTIONS:
Drug: VEDOLIZUMAB — Infusion at week 0 week 2 week 6 week 14 for all patients Infusion at week 22 for responder patient only
  Other Names: entyvio
Drug: ADALIMUMAB — For nonresponder patients only : Injection at week 22 week 24 week 26 and week 28
  Other Names: HUMIRA

SUMMARY:
The main objective of this project is to demonstrate the feasability of an endomicroscopic biomarker of efficacy of vedolizumab and adalimumab, in Ulcerative colitis (UC) by coupling vedolizumab to a fluorescent component, FITC (Fluorescein isothiocyanate) , and adalimumab to rhodamine.

This project should allow the development of a biomarker of therapeutic efficacy for vedolizumab and adalimumab that can be used in a single time-frame in vivo in humans, while respecting manufacturing standards and Good manufacturing procedures.

DETAILED DESCRIPTION:
Patients will be recruited before initiation of vedolizumab injections. The schedule for vedolizumab infusions will corresponding to the protocol follow-up visits (Week 0, W2, W6, W14, W22), and flexible sigmoidoscopy appointments will be performed at Week 0 and 22.

For responder patients, the end of the study will occured two weeks after the last vedolizumab infusion (W24).

At week 22, nonresponder patients to vedolizumab may be treated by adalimumab in the absence of contraindication and depending on the decision of the physician responsible for the patient. Patients will be treated every two weeks during 8 weeks. The protocol follow up will end 2 weeks after the fourth adalimumab injection.

During W0 and W22, colon biopsies will be collected. Blood samples will be collected on W0, W2, W6, W14, W22 (and W30 for non responder).

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe UC defined by an overall Mayo score ≥ 5 and an endoscopic sub-score ≥ 2 points and rectal bleeding score ≥ 1 point
* Extension > 15 cm from the anal margin
* Requiring treatment with biotherapy and meeting the indications for the treatment
* Affiliated with a social security scheme

Exclusion Criteria:

* Crohn's disease or unclassified colitis
* Severe acute colitis
* Requirement for immediate surgical treatment
* Previous treatment with vedolizumab or anti-TNF-α
* Contraindication to the use of vedolizumab or an anti-TNF-α agent
* Contraindication to the use of adalimumab
* Corticosteroid therapy > 20 mg/day
* Corticosteroid therapy started within the previous two weeks
* Conventional Immunosppressor started within the previous month
* Colonic dysplasia or known cancer
* Likelihood to refuse two rectosigmoidoscopies, performed eighteen weeks apart
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Demonstrate the feasibility of an ex vivo labeling of intestinal immune cells with a combination of two markers: vedolizumab-FITC and adalimumab-Alexa Fluor 647 | week 0
  Presence of fluorescent cells by Cellvizio® examination field for each of the antibodies: FITCcoupled vedolizumab and Alexa Fluor 647-coupled adalimumab at week 0 for all the patients.

SECONDARY OUTCOMES:
Quantify, ex vivo, the number of cells labeled with FITC-coupled vedolizumab in the intestinal mucosa of patients with moderate to severe UC that are associated with clinical remission at week 22 (W22) after the initiation of treatment with vedolizumab. | Week 22
  -Number of fluorescent cells by Cellvizio® examination field for each of the antibodies: FITC-coupled vedolizumab and Alexa Fluor 647-coupled adalimumab / Score of clinical response assessment
Evaluate the association between the number of cells labeled with FITC-coupled vedolizumab in the intestinal mucosa and the rate of clinical response induced by treatment with a standard dose of vedolizumab | week 22
  - Number of fluorescent cells / Mayo clinic sub-score
Evaluate the association between the number of cells labeled with FITC-coupled vedolizumab in the intestinal mucosa and the rate of endoscopic remission induced by treatment with a standard dose of vedolizumab | week 22
  - Number of fluorescent cells / Geboes sub-score
Evaluate the association between the number of cells labeled with FITC-coupled vedolizumab in the intestinal mucosa and the rate of histologic remission induced by treatment with a standard dose of vedolizumab | week 22
  - Number of fluorescent cells / Mayo endoscopic sub-score,
Evaluate the association between the number of cells labeled with FITC-coupled vedolizumab in the intestinal mucosa and the rate of clinical response induced by treatment with a standard dose of vedolizumab | week 22
  - Number of fluorescent cells / rectal bleeding score
Evaluate the association between the Alexa Fluor 647-coupled adalimumab biomarker, and the rate of clinical response at w30 to adalimumab | from week 0 to week 30
  Evolution of Number of fluorescent cells by Cellvizio® examination field for each of the antibodies between week 0 and week 22 / Mayo clinic sub-score
Evaluate the association between the Alexa Fluor 647-coupled adalimumab biomarker, and the rate of endoscopic remission at w30 to adalimumab | from week 0 to week 30
  Evolution of Number of fluorescent cells by Cellvizio® examination field for each of the antibodies between week 0 and week 22 / Mayo endoscopic sub-score,
Evaluate the association between the Alexa Fluor 647-coupled adalimumab biomarker, and the rate of endoscopic remission at w30 to adalimumab | from week 0 to week 30
  Evolution of Number of fluorescent cells by Cellvizio® examination field for each of the antibodies between week 0 and week 22 / Geboes sub-score
Evaluate the association between the Alexa Fluor 647-coupled adalimumab biomarker, and the rate of clinical remission at w30 to adalimumab | from week 0 to week 30
  Evolution of Number of fluorescent cells by Cellvizio® examination field for each of the antibodies between week 0 and week 22 / rectal bleeding score
Compare the number of positive immune cells FITC-coupled vedolizumab in the intestinal mucosa of patients with UC | week 0
  Average of Number of fluorescent cells FITC-coupled vedolizumab / patient
Compare the number of positive immune cells Alexa Fluor 647-coupled adalimumab in the intestinal mucosa of patients with UC | week 0
  Average of Number of fluorescent cells Alexa Fluor 647-coupled adalimumab/ patient

CONTACTS AND LOCATIONS:
Overall Officials: ARNAUD BOURREILLE, MD-PHD, Principal Investigator — Nantes University Hospital
Locations (4):
- France (4):
  - Chu Angers, Angers
  - Chd Vendee, La Roche-sur-Yon
  - Chu Nantes, Nantes
  - Chu Rennes, Rennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Queneherve L, Trang-Poisson C, Fantou A, Flamant M, Durand T, Bouguen G, Bregeon J, Oullier T, Amil M, Dewitte M, Bardot S, Blandin S, Braudeau C, Vibet MA, Josien R, Neunlist M, Bourreille A. Confocal laser endomicroscopy as predictive biomarker of clinical and endoscopic efficacy of vedolizumab in ulcerative colitis: The DETECT study. PLoS One. 2024 Apr 2;19(4):e0298313. doi: 10.1371/journal.pone.0298313. eCollection 2024. PMID 38564601